CLINICAL TRIAL: NCT07370571
Title: NO AXILLARY SURGERY IN EARLY BREAST CANCER
Brief Title: NO AXILLARY SURGERY IN EARLY BREAST CANCER (OXIGENATE)
Acronym: OXIGENATE
Status: Not yet recruiting | Type: Observational
Sponsor: Clinica Universidad de Navarra, Universidad de Navarra (Other)
Responsible Party: Principal Investigator, Isabel Rubio, MD, Clinica Universidad de Navarra, Universidad de Navarra
Other Study IDs: OXIGENATE
Record Dates: First submitted 2026-01-17; First posted 2026-01-27 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2025-11

CONDITIONS: Breast Cancer
Keywords: omission SLN, breast cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Early stage breast cancer ptients with omission of sentinel node biopsy
  Interventions: Procedure: Omission SLN

INTERVENTIONS:
Procedure: Omission SLN — Omission SLN

SUMMARY:
Prospective study will establish a comprehensive international registry specifically for patients who have undergone surgery for primary breast cancer without SLNB. The main objective of this registry is to gather detailed, real-world data on the outcomes of this particular treatment approach, providing insights into the clinical efficacy and quality of life of patients when SLNB is omitted.

DETAILED DESCRIPTION:
All patients with histologically confirmed invasive breast cancer and a negative axillary US who are candidates for omitting SLN biopsy or any axillary surgery will be informed about the possible participation in the study. The inclusion and exclusion criteria are verified by the investigator and written informed consent is obtained from the patient. Surgical treatment, pathological assessment and postoperative locoregional and systemic therapy should be conducted according to institutional and national standards. Since the OXYGENATE study in a non-interventional trial, the study sites do not deviate from their own institutional protocol at any timepoint. The follow up on patient status is conducted yearly during the first 5 years after surgery.

ELIGIBILITY:
Inclusion Criteria:

Older than 18 years old cT1-2 cN0 Negative preoperative assessment of the axilla Breast surgery as first treatment No axillary surgery Multifocal/ multicentric breast cancer Candidates to receive breast conserving surgery Written informed consent must be signed and dated by the patient and the investigator prior to inclusion.

Patients must be accessible for follow-up.

Exclusion Criteria Synchronous distant metastases Any axillary surgery Neoadjuvant treatment Previous malignancy Bilateral breast cancer Previous primary systemic therapy Pregnancy or breastfeeding Pre-operative diagnosis (cytology or histology) of axillary lymph node metastases Pre-operative radiological evidence of multiple involved or suspicious nodes Patients with psychiatric, addictive, or any disorder, which compromises their ability to give informed consent for participation in this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Early stage breast cancer patients with omission of SLN
Sampling Method: Probability Sample
Enrollment: 827 (Estimated)
Dates: Start 2026-03-01 (Estimated); Primary Completion 2027-03-30 (Estimated); Study Completion 2032-03-30 (Estimated)

PRIMARY OUTCOMES:
Axillary Recurrence | from enrollement to the end of follow up 5 years
  Determine the clinical efficacy of omitting a SLN i
3 year axillary recurrence | 3 years
  Identify if patients with no axillary surgery had an increased axillary recurrence

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF

DOCUMENTS (1):
  • Study Protocol (2025-06-20): https://cdn.clinicaltrials.gov/large-docs/71/NCT07370571/Prot_000.pdf